CLINICAL TRIAL: NCT03994705
Title: Phase I Safety Study of Descartes-11 in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Descartes-11 in Patients With Relapsed/Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Phase 1 enrollment completed. Further clinical development terminated.
Sponsor: Cartesian Therapeutics (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DC11A; 5R44CA221432-03 (NIH)
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
Keywords: CAR-T; CART; CAR T Cell; CAR T-Cell; Multiple Myeloma; BCMA; B cell maturation antigen; B-cell maturation antigen; Descartes-11
MeSH Terms: conditions — Multiple Myeloma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Level 1 (Experimental): Participants were administered Cyclophosphamide and Fludarabine for preconditioning on Days 1,2,3
  Participants were administered 10 million cells of Descartes-11 via intravenous catheter on Days 7,14
  Interventions: Biological: Descartes-11; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Level 2 (Experimental): Participants were administered Cyclophosphamide and Fludarabine for preconditioning on Days 1,2,3
  Participants were administered 32 million cells of Descartes-11 via intravenous catheter on Days 7,14
  Interventions: Biological: Descartes-11; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Level 3 (Experimental): Participants were administered Cyclophosphamide and Fludarabine for preconditioning on Days 1,2,3
  Participants were administered 100 million cells of Descartes-11 via intravenous catheter on Days 7,14
  Interventions: Biological: Descartes-11; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Level 4 A (Experimental): Participants were administered Cyclophosphamide and Fludarabine for preconditioning on Days 1,2,3
  Participants were administered 150 million cells of Descartes-11 via intravenous catheter on Days 7,14,21
  Interventions: Biological: Descartes-11; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Level 4B (Experimental): Participants were administered Cyclophosphamide and Fludarabine for preconditioning on Days 1,2,3
  Participants were administered 150 million cells of Descartes-11 via intravenous catheter on Days 7,10,14,21
  Interventions: Biological: Descartes-11; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Level 4C (Experimental): Participants were not administered Cyclophosphamide and Fludarabine for preconditioning on Days 1,2,3
  Participants were administered 150 million cells of Descartes-11 via intravenous catheter on Days 1,4, 7,10,14,21
  Interventions: Biological: Descartes-11

INTERVENTIONS:
Biological: Descartes-11 — CAR T-Cells
Drug: Fludarabine — Pre-conditioning chemotherapy
  Arms: Dose Level 1; Dose Level 2; Dose Level 3; Dose Level 4 A; Dose Level 4B
Drug: Cyclophosphamide — Pre-conditioning therapy
  Arms: Dose Level 1; Dose Level 2; Dose Level 3; Dose Level 4 A; Dose Level 4B

SUMMARY:
This Phase I study will test the safety and anti-myeloma activity of ascending doses of Descartes-11 (autologous CD8+ T-cells expressing an anti-BCMA chimeric antigen receptor) in eligible patients with active multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Active multiple myeloma that is refractory after at least 2 prior lines of therapy;
* measurable disease;
* adequate vital organ function; and
* no active infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-06-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Medical College of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Maus MV, Haas AR, Beatty GL, Albelda SM, Levine BL, Liu X, Zhao Y, Kalos M, June CH. T cells expressing chimeric antigen receptors can cause anaphylaxis in humans. Cancer Immunol Res. 2013 Jul;1(1):26-31. doi: 10.1158/2326-6066.CIR-13-0006. Epub 2013 Apr 7. PMID 24777247
- [Background] Beatty GL, Haas AR, Maus MV, Torigian DA, Soulen MC, Plesa G, Chew A, Zhao Y, Levine BL, Albelda SM, Kalos M, June CH. Mesothelin-specific chimeric antigen receptor mRNA-engineered T cells induce anti-tumor activity in solid malignancies. Cancer Immunol Res. 2014 Feb;2(2):112-20. doi: 10.1158/2326-6066.CIR-13-0170. PMID 24579088
- [Background] Teachey DT, Lacey SF, Shaw PA, Melenhorst JJ, Maude SL, Frey N, Pequignot E, Gonzalez VE, Chen F, Finklestein J, Barrett DM, Weiss SL, Fitzgerald JC, Berg RA, Aplenc R, Callahan C, Rheingold SR, Zheng Z, Rose-John S, White JC, Nazimuddin F, Wertheim G, Levine BL, June CH, Porter DL, Grupp SA. Identification of Predictive Biomarkers for Cytokine Release Syndrome after Chimeric Antigen Receptor T-cell Therapy for Acute Lymphoblastic Leukemia. Cancer Discov. 2016 Jun;6(6):664-79. doi: 10.1158/2159-8290.CD-16-0040. Epub 2016 Apr 13. PMID 27076371
- [Background] Lim WA, June CH. The Principles of Engineering Immune Cells to Treat Cancer. Cell. 2017 Feb 9;168(4):724-740. doi: 10.1016/j.cell.2017.01.016. PMID 28187291
- [Background] Brudno JN, Kochenderfer JN. Toxicities of chimeric antigen receptor T cells: recognition and management. Blood. 2016 Jun 30;127(26):3321-30. doi: 10.1182/blood-2016-04-703751. Epub 2016 May 20. PMID 27207799
- [Background] Ali SA, Shi V, Maric I, Wang M, Stroncek DF, Rose JJ, Brudno JN, Stetler-Stevenson M, Feldman SA, Hansen BG, Fellowes VS, Hakim FT, Gress RE, Kochenderfer JN. T cells expressing an anti-B-cell maturation antigen chimeric antigen receptor cause remissions of multiple myeloma. Blood. 2016 Sep 29;128(13):1688-700. doi: 10.1182/blood-2016-04-711903. Epub 2016 Jul 13. PMID 27412889
- [Background] GBD 2013 Mortality and Causes of Death Collaborators. Global, regional, and national age-sex specific all-cause and cause-specific mortality for 240 causes of death, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Jan 10;385(9963):117-71. doi: 10.1016/S0140-6736(14)61682-2. Epub 2014 Dec 18. PMID 25530442

RESULTS

PARTICIPANT FLOW:
Groups:
- Decartes-11 Dose Level 1: Participants were administered 10 million cells of Descartes-11 via intravenous catheter on Days 7, 14 Participants were administered cyclophosphamide and Fludarabine on Days 1,2,3
- Descates-11 Level 2: Participants were administered cyclophosphamide and Fludarabine for pre-conitioning on Days 1,2,3 Participants were administered 32 million cells of Descartes-11 via intravenous catheter on Days 7, 14
- Descartes-11 Dose Level 3: Participants were administered cyclophosphamide and Fludarabine for preconditioning on Days 1,2,3 Participants were administered 100 million cells of Descartes- 11 on Days 7,14
- Descartes-11 Dose Level 4A: Participants were administered Cyclophosphamide and Fludarabine for preconditioning on Days 1,2,3 Participants were administered 150 million cells of Descartes-11 via intravenous catheter on Days 7, 14,21
- Descartes-11 Dose Level 4B: Participants were administered Cyclophosphamide and Fludarabine for preconditioning on Days 1,2,3 Participants were administered 150 million cells of Descartes-11 via intravenous catheter on Days 7,10,14,17
- Descartes-11 Dose Level 4C: Participant did not receive preconditioning with cyclophosphamide or fludarabine, Participants were administered 150 million cells of Descartes-11 via intravenous catheter on Days 1,4,7,10,14,17
Period: Overall Study
Arm/Group | Decartes-11 Dose Level 1 | Descates-11 Level 2 | Descartes-11 Dose Level 3 | Descartes-11 Dose Level 4A | Descartes-11 Dose Level 4B | Descartes-11 Dose Level 4C
Started | 3 | 4 | 3 | 2 | 4 | 4
Completed | 3 | 4 | 3 | 2 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Level 1 Dose: 10 x 10^6 cells / kg
- Level 2 Dose: 32 x 10^6 cells / kg
- Level 3 Dose: 100 x 10^6 cells / kg
- Level 4A; Level 4B; Level 4C: 150 x 10^6 cells / kg
- Total: Total of all reporting groups
Arm/Group | Level 1 Dose | Level 2 Dose | Level 3 Dose | Level 4A | Level 4B | Level 4C | Total
Number analyzed (Participants) | 3 | 4 | 3 | 2 | 4 | 4 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 2 | 0 | 0 | 1 | 8
  >=65 years | 1 | 1 | 1 | 2 | 4 | 3 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 1 | 2 | 0 | 7
  Male | 2 | 2 | 2 | 1 | 2 | 4 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  White | 3 | 3 | 3 | 2 | 4 | 2 | 16
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Other-Non Hispanic | 0 | 0 | 0 | 0 | 0 | 1 | 1
  White (Hispanic) | 0 | 0 | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 3 | 2 | 4 | 4 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: Determine the safety of Descartes-11 in patients with relapsed/refractory multiple myeloma
Time Frame: Time Frame: 21 days
Population: Participants with treatment related adverse event
Measure: Count of Participants; unit: Participants
Groups:
- Dose-Escalation Level 1: Participants were administered Cyclophosphamide and Fludarabine for preconditioning
  Participants were administered 10 million cells of Descartes-11 via intravenous catheter
- Dose Level 2: Participants were administered Cyclophosphamide and Fludarabine for preconditioning
  Participants were administered 32 million cells of Descartes-11 via intravenous catheter
- Dose Level 3: Participants were administered Cyclophosphamide and Fludarabine for preconditioning
  Participants were administered 100 million cells of Descartes-11 via intravenous catheter
- Dose Level 4A; Dose Level 4B: Participants were administered Cyclophosphamide and Fludarabine for preconditioning
  Participants were administered 150 million cells of Descartes-11 via intravenous catheter
- Dose Level 4C: Participants were not administered Cyclophosphamide and Fludarabine for preconditioning
  Participants were administered 100 million cells of Descartes-11 via intravenous catheter
Arm/Group | Dose-Escalation Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4A | Dose Level 4B | Dose Level 4C
Number analyzed (Participants) | 3 | 4 | 3 | 2 | 4 | 4
Participants | 0 | 1 | 1 | 0 | 0 | 0

2. Secondary Outcome: Disease Assessment Based on International Myeloma Working Group (IMWG) Criteria
Description: Patience with Complete response (CR) according to the International Myeloma Working Group (IMWG).
Time Frame: Disease assessment is on Day 21 (or at least 14 days after first Descartes-11 infusion)
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-Escalation Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4A | Dose Level 4B | Dose Level 4C
Number analyzed (Participants) | 3 | 4 | 3 | 2 | 4 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Follow ups conducted on months 3,6,9,12.
Groups:
- Dose Level 4A: Participants were administered Cyclophosphamide and Fludarabine for preconditioning on Days 1,2,3
  Participants were administered 150 million cells of Descartes-11 via intravenous catheter on Days 7,14,21
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4A | Dose Level 4B | Dose Level 4C
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/4 | 0/3 | 0/2 | 0/4 | 1/4
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/4 | 1/3 | 1/2 | 1/4 | 0/4
Other Adverse Events (participants affected / at risk) | 3/3 | 2/4 | 2/3 | 1/2 | 3/4 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=4) | Dose Level 3 (N=3) | Dose Level 4A (N=2) | Dose Level 4B (N=4) | Dose Level 4C (N=4)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to Descartes-11
Febrile Neutropenia (Immune system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unlikely related to Desartes-11
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to Desartes-11
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to Desartes-11
Infusion reactions (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Related to Desartes-11
Plasmacytoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to Desartes-11
Dental Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to Desartes-11
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to Desartes-11
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to Desartes-11
Generalized weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to Desartes-11
Pathologic fractures of right femur and left humerus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to Desartes-11
Hypotension (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to Desartes-11
Hypoxia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to Desartes-11
Fever, etiology unknown (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to Desartes-11
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Unrelated to Desartes-11
Upper Resipratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to Desartes-11
Fever (preapheresis) (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Unrelated to Desartes-11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=4) | Dose Level 3 (N=3) | Dose Level 4A (N=2) | Dose Level 4B (N=4) | Dose Level 4C (N=4)
Aspartate aminotransferase increased (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Granulocyte count decreased (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Neutropenic fever (Immune system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (Etiology Unknown) (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion Related Reaction (Immune system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT03994705/Prot_SAP_000.pdf